CLINICAL TRIAL: NCT06887374
Title: Comparison of WHO Treatment of Acute Watery Diarrhea With or Without Probiotic (Bacillus Clausii) in Term of Mean Duration of Diarrhea in Children
Brief Title: Comparison of WHO Treatment of Acute Watery Diarrhea With or Without Probiotic (Bacillus Clausii) in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AWD-CH-LAHORE
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-03

CONDITIONS: Acute Watery Diarrhea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Patients received 2 billion spores of probiotic (Bacillus clausii) every 12 hours, contained in a small bottle along with standard treatment as per WHO guidelines.
  Interventions: Drug: Probiotic Bacillus Clausii
- No probiotic group (No Intervention): Patients received only standard treatment as per WHO guidelines.

INTERVENTIONS:
Drug: Probiotic Bacillus Clausii — Patients were given 2 billion spores of probiotic (Bacillus clausii) every12 hours, contained in a small bottle.
  Arms: Probiotic group

SUMMARY:
This study aimed to compare WHO treatment of acute watery diarrhea with or without probiotic (bacillus clausii) in term of mean duration of diarrhea in children

DETAILED DESCRIPTION:
Available literature regarding the use of probiotics is not conclusive and contains controversy, and local data is also scarce. Therefore, this study was planned to further explore the use of probiotics to furnish the local data. If significantly less mean duration of diarrhea is noted in the probiotic group, it will help to add probiotic bacillus clausii in routine treatment regimen recommended by WHO and to decrease costs associated with prolonged treatment. However, if otherwise results will be noted it will help to rule out use of probiotic bacillus clausii in children with acute diarrhea to avoid its unnecessary use.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Aged 6 to 59 months
* Suffering from acute watery diarrhea for ≤ 7 days

Exclusion Criteria:

* Children with blood in stool
* With prior antibiotics use
* Children under study with duration of stay more than 5 days
* clinical signs of a coexisting acute systemic illness like pneumonia, sepsis, meningitis, severely malnourished
* Immunocompromised children
* Hypersensitivity to probiotics
* With prior probiotic administration

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Stool frequency | 5 days
  A frequency of defecation of < 3 stools per day marked the effectiveness of the treatment.
Consistency of stools | 5 days
  The treatment was considered effective if the consistency of stools became semi-solid.

CONTACTS AND LOCATIONS:
Overall Officials: Talha Hassan, Principal Investigator — Children Hospital, Lahore, Pakistan; Muhammad Zeeshan, Study Director — Children Hospital, Lahore, Pakistan
Locations (1):
- Children Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.